CLINICAL TRIAL: NCT01877070
Title: Decision Making in Men With Early Stage Prostate Cancer Patients and Partners/Close Allies
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: 13-076
Record Dates: First submitted 2013-06-11; First posted 2013-06-13 (Estimated); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Low Risk Prostate Cancer
Keywords: assessments; 13-076

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

GROUPS / COHORTS (1):
- early stage prostate patients & their partners/close allies
  Interventions: Behavioral: assessments

INTERVENTIONS:
Behavioral: assessments

SUMMARY:
The purpose of this study is to collect information on how patients and their partners/close allies make treatment decisions when they have been diagnosed with early stage prostate cancer.

DETAILED DESCRIPTION:
Each patient and his partner will fill out assessments at baseline. Thereafter we will obtain the patients' treatment decision (AT or AS) within approximately 6 months. Once a patient makes a decision, he and his partner will complete another set of questionnaires. The patient and his partner will then complete the remaining questionnaires approximately 6, 12, 18, and 24 months following the treatment decision. We will examine the associations between baseline assessments , and the treatment decision as well as the changes in the assessments and the treatment decision. We will also assess associations between follow-up assessments and the decision to change a treatment decision from AS to AT. Data from patients and partners/close allies will generally be analyzed separately, thus patients who do not have a partner (or partner declines to participate) can still be enrolled and their psychosocial outcomes assessed.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Men who meet the NCCN guidelines for low risk prostate cancer, which include all of the following:

  * Most recent Gleason score ≤ 6, or clinical stage T1a or less;
  * Most recent PSA level below 10;
  * In the most recent biopsy, had fewer than 3 positive biopsy cores (with ≤ 50% cancer in each); OR the patient's doctor discussed active surveillance as a treatment option (as documented in visit notes of the patient's medical record)
* Are able to speak, read, write and understand English well enough to provide informed consent and complete study tasks
* Has not made a treatment decision prior to consent, as per self report
* 18 years of age or older

For partners/close allies:

* Considered a partner/close ally to the patient in the treatment making decision, as reported by the patient
* Are able to speak, read, write and understand English well enough to provide informed consent and complete study tasks
* 18 years old or older

Exclusion Criteria:

For patients:

* History of a cancer other than prostate cancer and non-melanoma skin cancer
* Significant psychiatric or cognitive disturbance sufficient, in the investigator's judgment, to preclude providing informed consent or participating in the study activities (i.e., acute psychiatric symptoms which require individual treatment)

For partners/close allies:

* Significant psychiatric or cognitive disturbance sufficient, in the investigator's judgment, to preclude providing informed consent or participating in the study activities (i.e., acute psychiatric symptoms which require individual treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from outpatient clinics at both the Urology Service at Memorial Sloan-Kettering Cancer Center (MSKCC). Patients may also be contacted by e-mail (securely using MSKSecure) or by mail.
Sampling Method: Non-Probability Sample
Enrollment: 541 (Estimated)
Dates: Start 2013-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
evaluate the impact of anxiety and the inability to tolerate ambiguity | 2 years
  on the decision making process in men with prostate cancer who are eligible for active surveillance and their partners/close allies. All participants will be administered a set of questionnaires that assess psychological and affective functioning, and treatment preferences.

SECONDARY OUTCOMES:
how partners/close allies influence the decision making process | 2 years
  participants will be administered a set of questionnaires that assess psychological and affective functioning, and treatment preferences.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/